CLINICAL TRIAL: NCT05272254
Title: Povidone Iodine Efficacy Study
Acronym: PIES
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Dorota Kopycka-Kedzierawski, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY00007064; 21-057-E (Other: Funder)
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Early Childhood Caries
MeSH Terms: interventions — Povidone-Iodine

STUDY DESIGN:
Intervention Model Description: At baseline, following oral rehabilitation in the operating room {10% (PVPI + Fluoride Varnish (FV)} will be compared to the current standard of care (Placebo + FV). Study participants will be followed for approximately 24 months post-baseline. The study interventions post-baseline will be administered at 3, 6, 9, 12, 15, 18, and 21 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Povidone Iodine (Experimental): 10% povidone iodine + fluoride varnish
  Interventions: Drug: 10% povidone iodine + FV
- Placebo (Placebo Comparator): Placebo (iced tea) + fluoride varnish
  Interventions: Other: Placebo +FV

INTERVENTIONS:
Drug: 10% povidone iodine + FV — applied to children's teeth
  Other Names: betadine
  Arms: Povidone Iodine
Other: Placebo +FV — applied to children's teeth
  Other Names: Iced tea
  Arms: Placebo

SUMMARY:
This is a single center, randomized, double-blind, placebo-controlled Phase II clinical trial (RCT) to evaluate the efficacy of topical 10% Polyvinylpyrrolidone-Iodine (PVPI) to prevent new cavitated caries lesions when applied to the teeth of children with Severe Early Childhood Caries (S-ECC). At baseline, following oral rehabilitation in the operating room {10% (PVPI + Fluoride Varnish (FV)} will be compared to the current standard of care (Placebo + FV). Study participants will be followed for approximately 24 months post-baseline. The study interventions post-baseline will be administered at 3, 6, 9, 12, 15, 18, and 21 months.

DETAILED DESCRIPTION:
Objectives:

Primary:

To assess the efficacy of 10% PVPI in children with S-ECC to prevent new cavitated caries lesions that require follow-up restorative/surgical intervention after oral rehabilitation in the Operating Room (OR) under general anesthesia.

The primary outcome variable is time from randomization to relapse. The development of an ICDAS caries code 3 (cavitated caries lesion) or higher lesion post dental surgery is the sentinel event to calculate time to relapse.

Secondary:

1. To determine incidence and severity of dental caries following oral rehabilitation in the OR.

   This outcome measure will be assessed by counting non-cavitated and cavitated carious lesions and any filled (due to caries), missing (due to caries) and sealed surfaces over the 2-year study period. The International Caries Diagnostic Assessment System (ICDAS) index will be used.
2. To determine diversity and composition of oral microbiota, including cariogenic Streptococcus Mutans, Lactobacilli and Candida species over the 2-year study period.

16S rRNA amplicon analysis of saliva from all participants will be used to identify bacterial taxa associated with dental caries. We will also quantify Colony Forming Units per mL (CFU/mL) of S. mutans, Lactobacilli and Candida species.

3. To determine the frequency of adverse event occurrence. Adverse events (AEs) will be collected from the parent/primary caregiver, as well as those observed by study investigators including unanticipated problems (UPs) and severe adverse events (SAEs) over the 2 year study period.

Population: Healthy children with S-ECC 24 to 71 months of age and their parents/primary caregivers from Rochester NY and the surrounding area will be invited to participate in this study. Enrolled children will be patients of record in the Pediatric Dentistry Division of the Eastman Institute for Oral Health (EIOH), University of Rochester, who require treatment for S-ECC in the OR under general anesthesia.

Phase or Stage: Phase II RCT Number of Sites: 1 site, University of Rochester Description of Intervention: The test agent will be 10% PVPI (Betadine Solution, Purdue Frederick Co., Stamford, CT). The placebo will consist of fluoride-free sterile water for injection USP and commercial powdered tea without sweetener or lemon (Lipton decaffeinated unsweetened tea, Lipton, Unilever, Englewood Cliffs, NJ) with addition of Red and Yellow Food Color (McCormick and Co., Inc., Hunt Valley, MD) to simulate the color of the 10% PVPI.

After drying the teeth, up to 15 µl of 10% PVPI or placebo solution will be applied to the child's teeth with a microbrush. Following application of the test agent (PVPI or placebo), FV (Duraflor®- 5% Sodium Fluoride Varnish, Bubble gum flavor, AMD Medicom, Inc. Quebec, Canada) that is the standard of care will be applied with the manufacturer's supplied applicator.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent/permission form
* Parents/primary caregivers willing to comply with all study procedures and be available for the duration of the study
* Male or female, of any race, ethnicity, aged 24 to 71 months and their parents/primary caregivers who are 18 years of age or older or emancipated minors
* In good general health as evidenced by medical history, per PI, and in compliance with current CDC, NYS Department of Health and URMC COVID-19 guidelines. American Society of Anesthesiologists (ASA) categories will be used; children classified as ASA I and ASA II will be eligible for the study.
* Diagnosed with Severe-Early Childhood Caries (S-ECC) requiring treatment in the operating room (OR). A diagnosis of S-ECC will be based on the definition in accordance with American Academy of Pediatric Dentistry (AAPD)

Exclusion Criteria:

* Having a known allergy or sensitivity to iodine or seafood, red or yellow food coloring, or to tea, including a hypersensitivity to fluoride varnish, or having thyroid disease, as determined by medical history
* Receiving or having received treatment with another investigational drug within 30 days of the baseline visit (V1)

Ages: 24 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 246 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Caries lesion | Randomization to relapse, up to 24 months
  The primary outcome variable is time from randomization to relapse. The development of an ICDAS caries code 3 (cavitated caries lesion) or higher lesion post dental surgery is the sentinel event to calculate time to relapse.

SECONDARY OUTCOMES:
Incidence and severity of dental caries | Randomization to relapse, up to 24 months
  To determine incidence and severity of dental caries following oral rehabilitation in the OR.
Diversity of oral microbiota | Randomization to relapse, up to 24 months
  To determine diversity of oral microbiota, including cariogenic Streptococcus Mutans, Lactobacilli and Candida species over the 2-year study period. Concentration (CFU/ml) will be measured
Adverse Event Occurrence | Enrollment to 24 months
  To determine the frequency of adverse event occurrence
Composition of Microbiota | Randomization to relapse, up to 24 months
  To determine composition of oral microbiota, including cariogenic Streptococcus Mutans, Lactobacilli and Candida species over the 2-year study period. Presence of species (yes or no) will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Dorota T Kopycka-Kedzierawski, DDS, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No